CLINICAL TRIAL: NCT01223391
Title: The Efficacy of Adjustable Lower Abdominal Compression in Neurogenic Orthostatic Hypotension
Brief Title: Abdominal Compression in Orthostatic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Jeffrey Basford, MD, PhD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-005203
Record Dates: First submitted 2010-09-28; First posted 2010-10-19 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Autonomic Failure; Orthostatic Hypotension
Keywords: orthostatic; abdominal compression
MeSH Terms: conditions — Pure Autonomic Failure; Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abdominal binder (Experimental): Standing with abdominal compression using elastic vs. non-elastic abdominal binders.
  Interventions: Other: Abdominal binder
- No abdominal binder (Placebo Comparator): Standing without abdominal compression
  Interventions: Other: No abdominal binder

INTERVENTIONS:
Other: Abdominal binder — External abdominal compression sequentially applied at 20 mmHg for 3 minutes, maximal tolerable level for 1.5 minutes and comfortable level for 2 minutes.
  Other Names: Elastic abdominal binder; Non-elastic abdominal binder
  Arms: Abdominal binder
Other: No abdominal binder — Standing without abdominal binder for 3 minutes
  Arms: No abdominal binder

SUMMARY:
The purpose of this study is to assess if abdominal binders that use pull strings to adjust compression (non-elastic) are more effective than standard elastic abdominal binders in attenuating neurogenic orthostatic hypotension.

DETAILED DESCRIPTION:
In 3 protocols, patients will undergo standing maneuvers, measured abdominal compressions, continuous BP monitoring and symptoms, ease-of-use and compliance scoring. In protocol 1, patients will exert abdominal compression to maximal tolerable and comfortable levels and values will be recorded. In protocol 2, patients will perform 3 standing maneuvers following a preceding rest period with and without abdominal compression at 20 mmHg (binders used in random order). In protocol 3, the standing maneuvers will be extended and the investigator will adjust binders to levels of abdominal compression corresponding to what patient gauged as maximal tolerable and comfortable levels. Comparison of outcome measures will establish which binder achieves higher abdominal compression, is easier to adjust, likely will be used in the future, if elastic and adjustable binders are equally effective in attenuating Orthostatic Hypotension and its associated symptoms at comparable pressures and which binder is more effective in recovering standing BP and improving orthostatic symptoms.

ELIGIBILITY:
SUBJECTS We will study 15 patients of both genders with neurogenic orthostatic hypotension (OH). Subjects will be recruited from the existing list of patients available in the database of the Autonomic Disorders Center.

Inclusion Criteria

1. Men and nonpregnant women aged 18-80 years.
2. Chronic neurologic conditions known to cause OH: multiple system atrophy (MSA), Parkinson's disease, autoimmune autonomic ganglionopathy or progressive autonomic neuropathy (e.g., diabetic, amyloid).
3. Orthostatic hypotension defined as a drop of systolic BP>30 mmHg or diastolic BP>15 mmHg.
4. Adrenergic failure of at least moderate severity defined as CASS-adrenergic ≥3.
5. Ambulatory and able to stand more than 3 minutes without pre-syncope.
6. BMI <29.
7. Ability to comply with study procedures and appointments.
8. Normal cognition (able to understand the study, learn the maneuvers, and follow complex commands).
9. Concomitant therapy with anticholinergic, alpha and beta agonists will be withdrawn 48 hours prior to autonomic evaluations. Midodrine will be withdrawn the night before evaluation. Fludrocortisone doses up to 0.2 mg per day will be permitted.

The diagnosis of probable MSA requires 1) the presence of orthostatic hypotension or urinary incontinence, and 2) poorly levodopa responsive parkinsonism or cerebellar ataxia.

The diagnosis of clinically definite Parkinson's disease requires 1) the presence of resting tremor, bradykinesia and rigidity, 2) clinical asymmetry, and 3) response to levodopa.

The diagnosis of autoimmune autonomic ganglionopathy requires 1) a sub-cute onset, 2) the presence of generalized and severe autonomic failure (CASS>6), 3) selective involvement of autonomic nerve fibers and 4) positive alpha-3 nicotinic acetylcholine receptor auto-antibodies.

Exclusion Criteria

1. Pregnant or lactating females.
2. Non-neurogenic OH, such as that due to medication or hypovolemia.
3. Chronic illnesses or other central nervous system conditions that affect autonomic function.
4. Established dementia.
5. Debilitating ataxia.
6. Moderate to severe lower extremity weakness.
7. Severe systemic illness, such as end-stage pulmonary, cardiac or renal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Difference between averaged standing blood pressure with and without binders | 3-7 minutes
  A 1-minute averaged blood pressure is measured at 3 minutes of standing without abdominal binder and at 3, 4.5 and 6.5 minutes of standing with abdominal binders. All measurements are obtained during a single session.

SECONDARY OUTCOMES:
Difference in orthostatic symptom score with and without binders | 3-7 minutes
  Orthostatic symptoms are measured at 3 minutes of standing without abdominal binder, and at 3, 4.5 and 6.5 minutes of standing with abdominal binders. All measurements are obtained during a single session.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Basford, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States